CLINICAL TRIAL: NCT00592566
Title: An Open Randomized Controlled Trial of Desmopressin, and Dexamethasone as Adjunctive Therapy in Patients With Pulmonary Hemorrhage Associated With Leptospirosis
Brief Title: Desmopressin and Dexamethasone Adjunctive Treatment for Leptospirosis
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Numbe of eligible patients has been decreased over time.
Sponsor: Mahidol University (Other)
Collaborators: Thailand Research Fund (Other)
Responsible Party: Prof. Yupin Suputtamongkol, Faculty of Medicine Siriraj Hospital, Mahidol University, Thailand
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DDP2003; RDG4630213
Record Dates: First submitted 2008-01-01; First posted 2008-01-14 (Estimated); Last update posted 2008-01-14 (Estimated); Status verified 2007-12

CONDITIONS: Leptospirosis
Keywords: Severe leptospirosis; Pulmonary hemorrhage
MeSH Terms: conditions — Leptospirosis | interventions — Dexamethasone; Deamino Arginine Vasopressin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (No Intervention): Standard supportive care
- 2 (Experimental): Dexamethasone treatment
  Interventions: Drug: Dexamethasone, desmopressin
- 3 (Experimental): Desmopressin treatment
  Interventions: Drug: Dexamethasone, desmopressin

INTERVENTIONS:
Drug: Dexamethasone, desmopressin — 200 mg of dexamethasone IV infusion OD for 3 days or 0.3 microgram/ kg of desmopressin in 50 ml of saline, as a 30- minute infusion
  Other Names: Minirin
  Arms: 2; 3

SUMMARY:
Background: Pulmonary involvement in leptospirosis has been reported to be on the increase and is emerging as the main cause of death due to leptospirosis in many countries, including Thailand.

Methods: A prospective randomized controlled trial of desmopressin or high dose dexamethasone as adjunctive therapy in patients with suspected pulmonary hemorrhage associated with leptospirosis was conducted between July 2003 and October 2006 at 5 hospitals in Thailand.

ELIGIBILITY:
Inclusion Criteria:

* adult patients (> 14 years) with suspected severe leptospirosis
* patients who presented with acute fever (oral temperature more than 38.00 C for <15 days) in the absence of an obvious focus of infection
* In the opinion of the attending physician might have pulmonary hemorrhage (i.e. history of hemoptysis, and/ or bilateral nodular or air space infiltration).

Exclusion Criteria:

* pregnant or breastfeeding
* those with history of bleeding disorder
* those who had underlying diseases such as chronic liver disease, diabetes mellitus
* those who received diuretic or glucocorticoid

Ages: 15 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2003-07; Primary Completion 2006-10 (Actual); Study Completion 2006-10 (Actual)

PRIMARY OUTCOMES:
Survival | during in hospital admission

SECONDARY OUTCOMES:
Days of mechanical ventilation | during hospital admission

CONTACTS AND LOCATIONS:
Overall Officials: Kanigar Niwattayakul, MD, Principal Investigator — Loei Hospital, Loei, Thailand:; Yupin Suputtamongkol, MD, Study Chair — Mahidol University
Locations (1):
- Loei Hospital, Mueng, Changwat Loei, Thailand